CLINICAL TRIAL: NCT02366390
Title: Efficacy of a Minimal Homebased Psychoeducative Intervention Versus Usual Care for the Management of Anxiety and Dyspnea in Patients With Severe Chronic Obstructive Pulmonary Disease
Brief Title: Dialogue Aimed at Reducing Anxiety in Patients With Severe COPD
Acronym: DIACOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DIACOL
Record Dates: First submitted 2015-02-06; First posted 2015-02-19 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Anxiety
Keywords: Psychoeducative; HADS; COPD; dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducative intervention (Experimental): A psychoeducative dialogue and one telephone booster session
  Interventions: Behavioral: Psychoeducative intervention
- Usual care (No Intervention): Usual care according to current guidelines.

INTERVENTIONS:
Behavioral: Psychoeducative intervention — Patient-education about feelings, cognitions, behaviors and bodily sensations related to management of dyspnea and associated anxiety
  Arms: Psychoeducative intervention

SUMMARY:
The purpose of this trial is to determine whether a minimal homebased psychoeducative intervention is effective in management of anxiety and dyspnea in patients with severe chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
In patients with severe chronic obstructive pulmonary disease (COPD) anxiety and dyspnea are described as the primary symptoms with a high impact on the patients quality of life and use of social services. Both pharmacological and non-pharmacological strategies aimed at reducing anxiety in patients with severe illness are challenged by low compliance and/or side-effect, which emphasized the need of focusing on treatment strategies that addresses the issues characteristic for a population with severe pulmonary disease.

The trial is a single-centre randomised clinical trial that test the hypothesis that a minimal homebased psychoeducative intervention reduces anxiety in patients with severe COPD. The primary outcome is anxiety assessed by the hospital and anxiety and depression scale (HADS), subscale for anxiety (HADS-A). Secondary outcomes are mastery of dyspnea measured by the Chronic Respiratory Questionnaire (CRQ), Health-related Quality of Life (HRQL) measured by the St. George Respiratory Questionnaire (SGRQ) and depression measured by the HADS, subscale for depression (HADS-D). The outcomes will be assessed at follow-up four weeks and three months after the intervention.

The trial population consist of patients with severe COPD affiliated the Department of Pulmonary & Infectious Diseases at Nordsjællands Hospital. Based on a sample size calculation sixty-six patients with severe COPD and associated anxiety will be randomised 1:1 to either intervention plus usual care or to usual care.

The intervention consist of a minimal psychoeducative dialogue delivered in the patient's home follow by a telephone booster session after two weeks. The intervention is based on a manual, where the theoretical foundation is cognitive behavior theory. The intervention is carried out by a nurse.

Our primary outcome of interest is intra-individual differences in HADS-A scores between baseline and last follow-up after three months. To analyse this with-in group difference in outcome we use paired t-test or Wilcoxon signed-rank. Differences between the groups will similarly be assessed with two-sample t-test or Wilcoxon rank-sum test. Same strategy will be used analyzing the secondary outcomes CRQ, SGRQ and HADS-D.

To include all points of follow-up and to evaluate the development with-in group and between groups we use a longitudinal regression model. Because of an expected high number of drop outs, the censuring due to death and missing data due to possibly lost to follow up will be handled appropriately, under supervision and in collaboration with an experienced bio-statistician. The sample size calculation is based on HADS-A, a paired design and a estimated drop-out of 33.3 %.

The trial is designed with the aim of giving nurses and other health professionals an instrument clinically applicable in proving care for patients with severe COPD and associated anxiety. Positive or negative results of the trial will be submitted to international journals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of COPD and classified as category C or D according to the Global initiative for Obstructive Lung Disease (GOLD), and who have a HADS - anxiety subscale score ≥ 8 and are willing to participate and able to provide written informed consent

Exclusion Criteria:

* Patients with a psychiatric diagnosis or pulmonary cancer or patients who are involved in any other interventional clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in HADS-A score from baseline to three months follow-up | Three months
  The Hospital Anxiety and Depression Scale (HADS), subscale for anxiety HADS-A is a self-completed questionnaire that measure symptoms of general anxiety

SECONDARY OUTCOMES:
Change in CRQ score from baseline to three months follow-up | Three months
  The Chronic Respiratory Questionnaire (CRQ) is a self-completed questionnaire measuring Health Related Quality of Life (HRQL) and mastery of dyspnea
Change in SGRQ score from baseline to three months follow-up | Three months
  The St. George´s Respiratory Questionnaire (SGRQ) is a self-completed questionnaire that measure HRQL
Change in HADS-D score from baseline to three months follow-up | Three months
  The Hospital Anxiety and Depression Scale (HADS), subscale for depression (HADS-D) ia a self-completed questionnaire that measure symptoms of general depression
Number of admissions | Three months
  Number of admission during the three months follow-up period
Length of Stay (LOS) | Three months
  Length of stay in hospitals during the three months follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Julie Midtgaard, PHD, Study Director — The University Hospital Centre for Health Research, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Nordsjællands Hospital, Department of Pulmonary & Infectious Diseases, Hillerød, Capital Region of Denmark, Denmark

REFERENCES:
- [Derived] Bove DG, Overgaard D, Lomborg K, Lindhardt BO, Midtgaard J. Efficacy of a minimal home-based psychoeducative intervention versus usual care for managing anxiety and dyspnoea in patients with severe chronic obstructive pulmonary disease: a randomised controlled trial protocol. BMJ Open. 2015 Jul 7;5(7):e008031. doi: 10.1136/bmjopen-2015-008031. PMID 26152326